CLINICAL TRIAL: NCT05484336
Title: Acute Effects of Three Doses of Spirulina in Glucose Beverages on Postprandial Glycemic Responses, Arterial Blood Pressure, and Subjective Appetite Responses: A Randomized Clinical Trial
Brief Title: Acute Effects of Spirulina on Postprandial Glycemic Responses and Arterial Blood Pressure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Agricultural University of Athens (Other)
Responsible Party: Principal Investigator, Aimilia Papakonstantinou, Assistant Professor in Nutrition and Metabolism, Agricultural University of Athens
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: HRBD 54 06/06/2022
Record Dates: First submitted 2022-07-30; First posted 2022-08-02 (Actual); Last update posted 2022-08-02 (Actual); Status verified 2022-07

CONDITIONS: Potential Abnormality of Glucose Tolerance; Appetitive Behavior; Blood Pressure
Keywords: blood glucose responses; blood pressure; spirulina; subjective appetite; blood glucose concentrations
MeSH Terms: conditions — Appetitive Behavior | interventions — Glucose

STUDY DESIGN:
Intervention Model Description: Crossover Assignment
Who Masked: Participant, Investigator
Masking Description: Double blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Glucose as reference food (Experimental): Thirteen healthy young adults, with BMI between 18 and 29.9 kg/m2 (male: 3, female:10) after 10-14h fast, consumed 50 g available carbohydrates from D-glucose, two times, in different weeks as reference food along with 300 mL water; and 50 g available carbohydrates from beverages containing 4, 6 and 8 g spirulina, tested once, in different visits, along with 300 mL water. There was a washout period of at least two days between visits. Fingertip capillary blood glucose samples were taken at 0, 15, 30, 45, 60, 90 and 120min postmeal. The first glucose sample was taken exactly 15min after the beginning of the consumption of the tested food.
  Interventions: Other: Glucose as reference food; Other: Beverage containing 4g spirulina; Other: Beverage containing 6g spirulina; Other: Beverage containing 8g spirulina
- Glucose beverage containing 4 g spirulina (Experimental): Thirteen healthy young adults, with BMI between 18 and 29.9 kg/m2 (male: 3, female:10) after 10-14h fast, consumed 50 g available carbohydrates from D-glucose, two times, in different weeks as reference food along with 300 mL water; and 50 g available carbohydrates from beverages containing 4, 6 and 8 g spirulina, tested once, in different visits, along with 300 mL water. There was a washout period of at least two days between visits. Fingertip capillary blood glucose samples were taken at 0, 15, 30, 45, 60, 90 and 120min postmeal. The first glucose sample was taken exactly 15min after the beginning of the consumption of the tested food.
  Interventions: Other: Glucose as reference food; Other: Beverage containing 4g spirulina; Other: Beverage containing 6g spirulina; Other: Beverage containing 8g spirulina
- Glucose beverage containing 6 g spirulina (Experimental): Thirteen healthy young adults, with BMI between 18 and 29.9 kg/m2 (male: 3, female:10) after 10-14h fast, consumed 50 g available carbohydrates from D-glucose, two times, in different weeks as reference food along with 300 mL water; and 50 g available carbohydrates from beverages containing 4, 6 and 8 g spirulina, tested once, in different visits, along with 300 mL water. There was a washout period of at least two days between visits. Fingertip capillary blood glucose samples were taken at 0, 15, 30, 45, 60, 90 and 120min postmeal. The first glucose sample was taken exactly 15min after the beginning of the consumption of the tested food.
  Interventions: Other: Glucose as reference food; Other: Beverage containing 4g spirulina; Other: Beverage containing 6g spirulina; Other: Beverage containing 8g spirulina
- Glucose beverage containing 8 g spirulina (Experimental): Thirteen healthy young adults, with BMI between 18 and 29.9 kg/m2 (male: 3, female:10) after 10-14h fast, consumed 50 g available carbohydrates from D-glucose, two times, in different weeks as reference food along with 300 mL water; and 50 g available carbohydrates from beverages containing 4, 6 and 8 g spirulina, tested once, in different visits, along with 300 mL water. There was a washout period of at least two days between visits. Fingertip capillary blood glucose samples were taken at 0, 15, 30, 45, 60, 90 and 120min postmeal. The first glucose sample was taken exactly 15min after the beginning of the consumption of the tested food.
  Interventions: Other: Glucose as reference food; Other: Beverage containing 4g spirulina; Other: Beverage containing 6g spirulina; Other: Beverage containing 8g spirulina

INTERVENTIONS:
Other: Glucose as reference food — Thirteen healthy, with BMI between 18 and 29.9 kg/m2 (male: 3, female:10) after 10-14h fast, consumed 50g glucose diluted in 250ml, tested two times, in different visits, within 5-10min. Fingertip capillary blood glucose samples were taken at baseline, 15, 30, 45, 60, 90 and 120min.
Other: Beverage containing 4g spirulina — Thirteen healthy, with BMI between 18 and 29.9 kg/m2 (male: 3, female:10) after 10-14h fast, consumed 50g glucose and 4g spirulina diluted in 250ml, tested once, within 5-10min. Fingertip capillary blood glucose samples were taken at baseline, 15, 30, 45, 60, 90 and 120min.
Other: Beverage containing 6g spirulina — Thirteen healthy, with BMI between 18 and 29.9 kg/m2 (male: 3, female:10) after 10-14h fast, consumed 50g glucose and 6g spirulina diluted in 250ml, tested once, within 5-10min. Fingertip capillary blood glucose samples were taken at baseline, 15, 30, 45, 60, 90 and 120min.
Other: Beverage containing 8g spirulina — Thirteen healthy, with BMI between 18 and 29.9 kg/m2 (male: 3, female:10) after 10-14h fast, consumed 50g glucose and 8g spirulina diluted in 250ml, tested once, within 5-10min. Fingertip capillary blood glucose samples were taken at baseline, 15, 30, 45, 60, 90 and 120min.

SUMMARY:
This study investigated the effects of three doses of spirulina in glucose beverages on postprandial glycemic responses, arterial blood pressure, and subjective satiety.

DETAILED DESCRIPTION:
This study aimed to determine the effects of three different doses (4, 6 and 8 g) of spirulina in glucose beverages on postprandial glycemic responses, blood pressure, and subjective appetite responses in healthy young adults.

ELIGIBILITY:
Inclusion Criteria:

* healthy
* non-smokers
* men and women
* body mass index between 18 and 24.9 kg/m2
* normal blood pressure (systolic blood pressure <120 mmHg and diastolic blood pressure <80 mmHg)
* normal fasting blood glucose concentrations (<100 mg/dL)

Exclusion Criteria:

* Medical conditions (e.g., cardiovascular diseases, diabetes mellitus, kidney or liver conditions, severe clinical depression, gastrointestinal disorders)
* Under medications known to affect glycemia (glucocorticoids, metformin, thiazide diuretics)
* Allergy to spirulina
* Pregnancy
* Lactation
* Competitive sports
* Alcohol abuse
* Drug dependency

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 13 (Actual)
Dates: Start 2022-06-07 (Actual); Primary Completion 2022-07-15 (Actual); Study Completion 2022-07-26 (Actual)

PRIMARY OUTCOMES:
Capillary blood glucose responses | 2 hours
  Clinically useful change in blood glucose, defined as the restoration of glucose within normal limits during 2hr glucose tolerance test
Blood pressure | 2 hours
  Useful change in systolic and diastolic blood pressure before and 2hr after consumption of the three doses of spirulina in beverages

SECONDARY OUTCOMES:
Subjective appetite ratings | 2 hours
  Useful change in subjective appetite using visual analogue scales with a score 0 to 10 (given in form of booklet, one scale per page) at baseline, 15, 30, 45, 60, 90 and 120. The minimum or maximum score will be evaluated if it is better or worse depending on the appetite variable e.g. hunger, satiety, desire to eat etc.

CONTACTS AND LOCATIONS:
Overall Officials: Emilia Papakonstantinou, PhD, Principal Investigator — Agricultural University of Athens
Locations (1):
- Agricultural University of Athens, Athens, Attica, Greece

IPD SHARING:
Plan to Share IPD: No